CLINICAL TRIAL: NCT05763056
Title: Comparison of the Effects of Intubation With a Machintosh Laryngoscope, McGrath Videolaryngoscope and C-Mac Videolaryngoscope on Intra-ocular Pressure, Optic Nerve Sheath Diameter and Haemodynamic Parameters
Brief Title: Effects of Intubation on Intra-ocular Pressure and Optic Nerve Sheath Diameter
Acronym: [Intubation]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Erol Karaaslan, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ekaraaslan4
Record Dates: First submitted 2023-01-17; First posted 2023-03-10 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Intraocular Pressure
Keywords: laryngoscope; intraocular pressure; optic nerve sheath

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective Randomized, Placebo-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- McGrath videolaryngoscopy (Active Comparator): It is a portable videoryngoscope weighing only 325 grams. The CameraStickTM component consists of a light source and a miniature camera, and the image is displayed on a 1.7 inch LCD (Liquid Crystal Display) screen mounted on top of the laryngoscope handle. At the same time, the LCD screen maintains visual contact with the patient and the laryngoscope, can be rotated up to 90°, allowing the user to work in a comfortable posture while performing tracheal intubation. The blade length is suitable for children over 5 years old and adults, thus reducing the trouble of storing different sized blades in the emergency intubation trolley. The blades are sterile and there is no risk of contamination as they are disposable.
  Interventions: Procedure: McGrath videolaryngoscopy; Procedure: C-MAC videolaryngoscopy; Device: Direct laryngoscopy
- C-MAC videolaryngoscopy (Active Comparator): Considering the importance of first attempt success in intubation, their use in emergency airway management has increased due to the high first attempt success rate in C-MAC VLs. In patients with cervical spine injury, semi-rigid collars used to prevent neck extension and neck movements cause poor laryngeal vision with Direct laryngoscope and difficulty intubation. C-MAC Video laryngoscope provides a better laryngeal view in these patients
  Interventions: Procedure: McGrath videolaryngoscopy; Procedure: C-MAC videolaryngoscopy; Device: Direct laryngoscopy
- Direct laryngoscopy (Active Comparator): Macintosh laryngoscopy is still one of the most commonly used advanced airway methods today. For an ideal glottis view in direct laryngoscopy, the mouth and larynx should be in alignment. For this, longitudinal flexion and head extension maneuvers are performed. Reasons such as the clinical situation during intubation and the anatomical variation in the patient may prevent this maneuver from being performed.
  Interventions: Procedure: McGrath videolaryngoscopy; Procedure: C-MAC videolaryngoscopy; Device: Direct laryngoscopy

INTERVENTIONS:
Procedure: McGrath videolaryngoscopy — The McGrath video laryngoscope has a thin, disposable, clear, regularly shaped blade similar to a Macintosh blade and a large LCD display attached to the arm. It is lighter in weight and the Mc VL has a small camera at the tip, with a more compact screen and handle that can make tracheal intubation easier and faster in normal or difficult airway. The smaller volume, thinner and portrait screen helps reduce blind spots
Procedure: C-MAC videolaryngoscopy — The Macintosh blade is attached to the handle and the light beam is passed through the blade tip into a small metal guide tube indented 40 mm. The camera cable is connected to the control unit and the optical cable is connected to the light source. The video macintosh system is installed in a small trolley for easy portability of the device. The trolley supports an 8-inch monitor mounted on a rotating arm on the patient's left side. C-MAC VL devices can create continuous video recordings or static images on a secure removable digital card. The electronic module includes 2 buttons for photo and video shooting. In addition, the image of the C-MAC VL device can be viewed on other devices or recorded via a standard video output port. 3 C-MAC VL reusable metal macintosh blades (sizes 2 to 4) can be used for adult patients. These non-disposable knives have a closed design without gaps in terms of hygiene and have beveled edges to prevent tissue damage.
Device: Direct laryngoscopy — During intubation with a direct laryngoscope (DL), the laryngoscope is inserted into the oral cavity from the right side of the mouth, the tongue is pushed to the left, and after advancing up to the vallecula, it hangs up and forward. In this way, the floor of the mouth and the epiglottis structure are removed from the field of view. If a straight blade laryngoscope is to be used, it is advanced so that the epiglottis remains under the blade after viewing the epiglottis (1). In DL, manipulations such as head extension, sniffing position, and compression of the cricoid cartilage may be required to facilitate visualization of the vocal folds. In 10-15% of the complications experienced during intubation with DL, there are problems related to the angle of view.

SUMMARY:
Brief Summary:

In this study, the investigators aimed to compare the effects of different types of endotracheal instruments (Machintosh laryngoscope, McGrath videoingoscope and C-Mac videoryngoscope) on intraocular pressure, optic nerve diameter and hemodynamic parameters.

DETAILED DESCRIPTION:
Detailed Description:

Laryngoscopy and endotracheal intubation cause increased intracranial pressure due to hypoxia, hypercapnia, straining, or coughing. It may be an indirect result of increased arterial and venous pressure, as well as a direct effect of intubation.

With the emergence of neuroimaging techniques and new diagnostic tools, various methods have been developed that can replace invasive methods, which are the gold standard in intraocular pressure measurement. However, invasive methods such as intraventricular and intraparenchymal catheter systems have some disadvantages and are associated with significant risks in terms of infection, bleeding, and time lost until follow-up.

The intraorbital subarachnoid space surrounding the optic nerve shows the same pressure variation as the intracranial subarachnoid space, and any increase in intracranial pressure is also seen in the orbital subarachnoid space. With the increase in intracranial pressure, the optic nerve, optic nerve sheath diameter, and subarachnoid space enlarge. There are many studies reporting that optic nerve sheath diameter can be evaluated using ultrasonography. Although there is no clear cut-off value for optic nerve sheath diameter, previous studies have found that an optic nerve sheath diameter of 5.0 mm and above may indicate an increase in intracranial pressure.

Previous studies have determined that the distribution of intraocular pressure in the adult population varies between 11 mmHg and 21 mmHg, and the mean intraocular pressure is 16.5 mmHg. It is well known that the sympathoadrenergic response caused by laryngoscopy and tracheal intubation significantly increases intraocular pressure (at least 10-20 mmHg). In addition, intravenous pressure and intraocular pressure increase due to cough, airway obstruction, succinylcholine use, hypoxia and hypercapnia during intubation.

In this study, the investigators aimed to compare the effects of different types of endotracheal instruments (Machintosh laryngoscope, McGrath videoingoscope and C-Mac videoringoscope) on intraocular pressure, optic nerve sheath diameter and hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Non-ophthalmic surgery
* Mallampati I or II classifications
* American Society of Anesthesiologists (ASA) I-II

Exclusion Criteria:

* Glaucoma,
* Diabetes mellitus,
* Cardiovascular diseases,
* Pulmonary diseases,
* ASA 3 and 4
* Body Mass Index (BMI) greater than 30
* Eye surgery
* Difficult intubation (Mallampati score of 3 or 4, thyromental distance of less than 6 cm and a maximum mouth opening of less than 3 cm)
* Intraocular pressure value more than 20 mmHg
* More than two intubation attempts
* A risk of regurgitation patients
* History of obstetric surgery
* Allergies to propofol, fentanyl or rocuronium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure-1 | Intraocular pressure will be measured at before induction
  Right and left intraocular pressures will be measured with a Tono-pen (AVIA) (Reichert Technologies, Depew, NY, USA) device by an ophthalmologist unaware of the patient group. Initial intraocular pressure value will measured without using any sedative drugs. An ophthalmologist, unaware of the randomization, measured intraocular pressure using ocular sonography. It will be measured as intraocular pressure: mmHg.
Intraocular pressure-2 | Intraocular pressure will be measured at just before laryngoscopy and intubation
  Right and left intraocular pressures will be measured with a Tono-pen (AVIA) (Reichert Technologies, Depew, NY, USA) device by an ophthalmologist unaware of the patient group. Initial intraocular pressure value will measured without using any sedative drugs. An ophthalmologist, unaware of the randomization, measured intraocular pressure using ocular sonography. It will be measured as intraocular pressure: mmHg.
Intraocular pressure-3 | Intraocular pressure will be measured at immediately after intubation
  Right and left intraocular pressures will be measured with a Tono-pen (AVIA) (Reichert Technologies, Depew, NY, USA) device by an ophthalmologist unaware of the patient group. Initial intraocular pressure value will measured without using any sedative drugs. An ophthalmologist, unaware of the randomization, measured intraocular pressure using ocular sonography. It will be measured as intraocular pressure: mmHg.
Intraocular pressure-4 | Intraocular pressure will be measured at 5 minutes after intubation
  Right and left intraocular pressures will be measured with a Tono-pen (AVIA) (Reichert Technologies, Depew, NY, USA) device by an ophthalmologist unaware of the patient group. Initial intraocular pressure value will measured without using any sedative drugs. An ophthalmologist, unaware of the randomization, measured intraocular pressure using ocular sonography. It will be measured as intraocular pressure: mmHg.
Intraocular pressure-5 | Intraocular pressure will be measured at 10 minutes after intubation
  Right and left intraocular pressures will be measured with a Tono-pen (AVIA) (Reichert Technologies, Depew, NY, USA) device by an ophthalmologist unaware of the patient group. Initial intraocular pressure value will measured without using any sedative drugs. An ophthalmologist, unaware of the randomization, measured intraocular pressure using ocular sonography. It will be measured as intraocular pressure: mmHg.

SECONDARY OUTCOMES:
Optic nerve diameter measurement-1 | Optic nerve diameter measurement-1 will be measured at before induction
  Optic nerve diameter measurements will be made from the transverse and sagittal planes of both eyes using a linear 6-12 MHz transducer (EsaoteMyLabFive, Genoa, Italy). An ophthalmologist, unaware of the randomization, measured optic nerve diameter using ocular sonography. It will be measured as optic nerve sheath diameter: mm.
Optic nerve diameter measurement-2 | Optic nerve diameter measurement-2 will be measured at just before laryngoscopy and intubation
  Optic nerve diameter measurements will be made from the transverse and sagittal planes of both eyes using a linear 6-12 MHz transducer (EsaoteMyLabFive, Genoa, Italy). An ophthalmologist, unaware of the randomization, measured optic nerve diameter using ocular sonography. It will be measured as optic nerve sheath diameter: mm.
Optic nerve diameter measurement-3 | Optic nerve diameter measurement-3 will be measured at immediately after intubation
  Optic nerve diameter measurements will be made from the transverse and sagittal planes of both eyes using a linear 6-12 MHz transducer (EsaoteMyLabFive, Genoa, Italy). An ophthalmologist, unaware of the randomization, measured optic nerve diameter using ocular sonography. It will be measured as optic nerve sheath diameter: mm.
Optic nerve diameter measurement-4 | Optic nerve diameter measurement-4 will be measured at 5 minutes after intubation
  Optic nerve diameter measurements will be made from the transverse and sagittal planes of both eyes using a linear 6-12 MHz transducer (EsaoteMyLabFive, Genoa, Italy). An ophthalmologist, unaware of the randomization, measured optic nerve diameter using ocular sonography. It will be measured as optic nerve sheath diameter: mm.
Optic nerve diameter measurement-5 | Optic nerve diameter measurement-5 will be measured at 10 minutes after intubation
  Optic nerve diameter measurements will be made from the transverse and sagittal planes of both eyes using a linear 6-12 MHz transducer (EsaoteMyLabFive, Genoa, Italy). An ophthalmologist, unaware of the randomization, measured optic nerve diameter using ocular sonography. It will be measured as optic nerve sheath diameter: mm.

CONTACTS AND LOCATIONS:
Overall Officials: Erol Karaaslan, assoc prof, Study Director — Inonu University Medical Faculty , malatya.turkey
Locations (1):
- Inonu University Medical Faculty, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900